CLINICAL TRIAL: NCT02624466
Title: Part 1 of: 'Conceptualisation and Validation of a Paradigm Based on Uraemic Toxins for Management of Chronic Kidney Disease in Paediatric Patients (UToPaed)'
Brief Title: Uraemic Toxins in Chronic Kidney Disease Paediatric Patients: Observational Study
Acronym: UToPaed_1
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor
Other Study IDs: UGent_UToPaed_1
Record Dates: First submitted 2015-11-16; First posted 2015-12-08 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Disease
Keywords: Pediatrics; Nephrology; Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CKD - no dialysis: Follow-up of CKD progress by frequent assessment of: concentration of uraemic toxins in blood, anthropometry, cardio-vascular parameters, body composition monitoring, dietary assessment, psycho-social questionnaires, sleep disorders, stool, nails.
  Interventions: Other: CKD progress
- Patients on PD: Follow-up of CKD progress by frequent assessment of: concentration of uraemic toxins in blood, urine and PD fluid, anthropometry, cardio-vascular parameters, body composition monitoring, dietary assessment, psycho-social questionnaires, sleep disorders, stool, nails.
  Interventions: Other: CKD progress
- Patients on HD: Follow-up of CKD progress by frequent assessment of: concentration of uraemic toxins in blood, urine and spent dialysate, anthropometry, cardio-vascular parameters, body composition monitoring, dietary assessment, psycho-social questionnaires, sleep disorders, stool, nails.
  Interventions: Other: CKD progress

INTERVENTIONS:
Other: CKD progress — CKD progress

SUMMARY:
Children with chronic kidney disease (CKD) suffer from one of the most devastating diseases in childhood resulting in a lifelong need for health care, and a 3 times decreased life expectancy. In addition, they have important comorbidities that negatively impact on their quality of life and integration in society, jeopardizing their future even after a potential transplantation. Retention of uraemic toxins is accepted to play a major role in the pathogenesis of the comorbid conditions, but studies in children are lacking. Furthermore, there are currently no good tools to evaluate severity and monitor adequacy of treatment, resulting in suboptimal management.

The overall scientific objective of this four years UToPaed IWT-TBM project is to provide the clinician with new diagnostic and therapeutic tools for the management of children with CKD, based on the improved understanding of uraemic toxicity.

In this first part of UToPaed, the investigators will associate concentrations of a wide variety of uraemic toxins with different comorbidities in CKD children, i.e. growth, protein-energy wasting, quality of life, cardiovascular risk factors, circadian rhythm, sleep quality, and psychosocial and neurocognitive functioning (i.e. cross-sectional and longitudinal). The toxins of which concentrations are best correlated with comorbidities during the progress of CKD and eventually have representative kinetics (UToPaed - part 2: Kinetic analysis) will be selected as markers. These markers will be, together with the comorbidities, further tracked after interventions, i.e. starting on dialysis, transplantation, changes in dialysis strategy (UToPaed - part 3 - intervention study).

From the validated kinetic models (UToPaed - part 2 and 3), an open access user-friendly prediction simulator (PAEDSIM) based on patient characteristics and marker concentrations will be developed to optimise and individualise the dialysis therapy.

By providing clinicians with more advanced and appropriate tools to improve management of all children with CKD, i.e. better assessment of the degree of renal dysfunction, better determination of the ideal time to start renal replacement therapy, and more accurate monitoring of dialysis adequacy, the investigators aim to improve neurocognitive and psychosocial functioning (short term), growth, maturation into puberty, and social integration (median term) and survival (long term).

DETAILED DESCRIPTION:
This is a prospective observational multicenter study in children (≤ 18 years) with chronic kidney disease (CKD) stage 2 to 5D with or without renal replacement therapy. In this study, 60 children with CKD stage 2 - 5 (without renal replacement therapy)(GROUP 1), 30 children with CKD stage 5D treated with peritoneal dialysis (GROUP 2) and 30 children with CKD stage 5D treated with haemodialysis (GROUP 3) will be followed for a total duration of 24 months.

The study participants are evaluated on their standard visit at the outpatient clinic every 3 months. At this visit, a blood sample for uraemic toxin concentration is withdrawn and several co-morbidities (growth, protein-energy wasting, cardiovascular disease, quality of life, psychosocial functioning, sleep, attention and executive functions) are assessed. Anthropometric parameters, dietary assessment, stool evaluation, nail evaluation, office and 24 hours ambulatory blood pressure monitoring, echocardiography and questionnaires are used to map out the several co-morbidities.

Blood analyses are performed to get the concentrations of a wide variety of uraemic toxins: i.e. small water soluble solutes, middle molecules and protein-bound solutes. All blood analyses within this project are performed in the Ghent University Hospital: i.e. urea, creatinine, calcium, and phosphorus are determined in the routine laboratory of the Ghent University Hospital using standard methods, while all other uraemic toxins are determined in the laboratory of the Nephrology Section using ELISA and (in-house developed) HPLC/UPLC techniques. For the protein-bound solutes two runs are needed to distinguish between total and free fractions of the protein-bound solutes.

The following actions are performed prior to enrolment:

* Review medical history to determine eligibility based on inclusion/exclusion criteria
* Obtain document consent from participant (>12 years) and parent/representative on study consent form
* Schedule study visits for individuals who are eligible and available for the duration of the study
* Provide potential participants with instructions needed to prepare for first study visit

Baseline visit:

* Verify inclusion/exclusion criteria.
* Obtain and record general patient information: age, sex, medical history, underlying kidney disease, medication history, current medication chart, dialysis settings and demographic information
* Assessment of dietary assessment by a skilled dietician by means of 3-day diet diary or three 24-hours recall
* Perform clinical assessment including anthropometric parameters and office blood pressure
* Perform a body composition monitoring (BCM) in children > 10 kg
* Collection of blood sample (all groups; EDTA immediately on ice; serum 15-30 minutes rest and subsequently on ice), 24 hours urine sample (group 2; 24 hours prior to visit), intradialytic urine sample (group 3) and 24 hours dialysate collection (group 2; 24 hours prior to visit) for determination of uraemic toxin concentration

Intermediate visits:

* Obtain general patient information: medication chart, changes in medical situation and dialysis settings
* Assessment of dietary intake by a skilled dietician by means of 3-day diet diary or three 24-hours recall every 3 months
* Perform clinical assessment including anthropometric parameters and office blood pressure
* Perform BCM 3-monthly in children > 10 kg with renal replacement therapy (group 2 and 3) and 1-yearly in children > 10 kg without renal replacement therapy (group 1)
* Collection of blood sample (group 1 to 3; EDTA immediately on ice; serum 15-30 minutes rest and subsequently on ice), 24 hours urine sample (group 2 and 3; 24 hours prior to visit) and 24 hours dialysate collection (group 2; 24 hours prior to visit) every 3 months for determination of uraemic toxin concentration.
* Collection of stool sample for determination of microbiota and metabolome 1-yearly (only participants of Ghent University Hospital)
* Collection of nails for determination of carbamylation process every 6 months (only participants of Ghent University Hospital)
* Perform echocardiography by a skilled paediatric cardiologist every year (visit 2, 5)
* Withdraw questionnaires from the parent and/or child assessing quality of life, attention, sleep, executive function and parental functioning every 6 months (visit 2, 4, 6, 8)
* Perform 24 hours ambulatory blood pressure measurement in children > 6 years once a year (visit 2, 5)

Final Study Visit:

* Obtain general patient information: medication chart, changes in medical situation and dialysis settings (detailed overview appendix 2)
* Assessment of dietary assessment by a skilled dietician by means of 3-day diet diary or three 24-hours recall
* Perform clinical assessment including anthropometric parameters and office blood pressure
* Perform a body composition monitoring (BCM) in children > 10 kg
* Collection of blood sample (group 1 to 3; EDTA immediately on ice; serum 15-30 minutes rest and subsequently on ice), 24 hours urine sample (group 2 and 3; 24 hours prior to visit) and 24 hours dialysate collection (group 2; 24 hours prior to visit) for determination of uraemic toxin concentration
* Perform echocardiography by a skilled paediatric cardiologist
* Perform 24 hours ambulatory blood pressure measurement in children > 6 years

The following socio-demographic questionnaires are asked to be completed:

1. Assessment of quality of life (QoL)

   * PedsQL for children (5-18 years)
   * PedsQL for children, disease specific (8-12 years, 13-18 years)
   * Parent Proxy Report by parents (2-4 years, 5-7 years, 8-12 years, 13-18 years)
   * Parent Proxy Report, disease specific by parents (8-12 years, 13-18 years)
2. Assessment of psychological wellbeing

   * YSR for children (> 11 years)
   * CBCL/TRF by parent/teachers (1,5-5 years, 6-18 years)
   * CBSK for children (8-12 years), CBSA for children (13-18 years)
3. Assessment of attention & executive functions

   * DBDRS by parents, teachers (6-16 years)
   * BRIEF by parents/teachers (5-18 years)
4. Assessment of sleep

   * ESS questionnaire by parents
   * CSHQ questionnaire by parents
5. Assessment of family functioning

   * PIP by parents
   * HADS by parents
   * PSI-S by parents
   * PPS by parents
   * CVS by parents

ELIGIBILITY:
Subject Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged ≤ 18 years
* Diagnosed with chronic kidney disease stage 2 to 5D, according to the K/DOQI guidelines.

Subject Exclusion Criteria:

* Partially exclusion of children and/or parents who cannot fill in the questionnaires due to language barriers. They will be excluded only from the questionnaires; the other comorbidities will be followed.
* Partially exclusion of children who cannot fill in the questionnaires due to mental retardation. They will be excluded only from the questionnaires; the other comorbidities will be followed.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: CKD patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-10; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Detect whether uraemic toxin concentrations are correlated with the different measured co-morbidities | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Eloot, Prof Dr, Principal Investigator — Ghent University Hospital - Nephrology; Johan Vande Walle, Prof Dr, Study Chair — Ghent University Hospital - Paediatric Nephrology; Ann Raes, Prof Dr, Study Chair — Ghent University Hospital - Paediatric Nephrology; Wim Van Biesen, Prof Dr, Study Chair — Ghent University Hospital - Nephrology; Evelien Snauwaert, Study Chair — Ghent University Hospital - Paediatric Nephrology
Locations (1):
- Ghent University Hospital - Nephrology, Ghent, Belgium